CLINICAL TRIAL: NCT06070701
Title: NOL-Guided Superficial Parasternal Intercostal Plane Block Versus Erector Spinae Plane Block in Open Heart Surgery With Cardiopulmonary Bypass - A Propensity Matched Non-Inferiority Clinical Trial
Brief Title: NOL-Guided Superficial Parasternal Intercostal Plane Block Versus Erector Spinae Plane Block
Acronym: NESP-II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institutul de Urgenţă pentru Boli Cardiovasculare Prof.Dr. C.C. Iliescu (Other)
Responsible Party: Principal Investigator, Balan Ion Cosmin, Principal Investigator, Institutul de Urgenţă pentru Boli Cardiovasculare Prof.Dr. C.C. Iliescu
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21330
Record Dates: First submitted 2023-09-22; First posted 2023-10-06 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Analgesia
Keywords: cardiac surgery; regional anesthesia; nociception; enhanced rehabilitation; erector spinae plane block; superficial parasternal intercostal plane block
MeSH Terms: conditions — Agnosia | interventions — Anesthetics, General; Morphine

STUDY DESIGN:
Intervention Model Description: Propensity score matching
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SUPERFICIAL PARASTERNAL INTERCOSTAL PLANE BLOCK (SPIPB) (Experimental): Following induction, ropivacaine 0.5% (1.5 mg/kg per each side) with dexamethasone 8mg/20ml is deposited under ultrasound guidance in the plane between the intercostal muscles and the pectoralis major muscles, targeting the anterior cutaneous branches of the intercostal nerves.
  Interventions: Procedure: Superficial Parasternal Block (SIPB); Drug: General anesthetic; Drug: Morphine
- ERECTOR SPINAE PLANE BLOCK (ESPB) (Active Comparator): Before induction, ropivacaine 0.5% (1.5 mg/kg per each side) with dexamethasone 8mg/20ml is deposited under ultrasound guidance between the transverse process of the 5th thoracic vertebra and the erector spinae muscle, targeting the dorsal and ventral rami of the spinal nerves.
  Interventions: Procedure: Erector Spinae Plane Block (ESPB); Drug: General anesthetic; Drug: Morphine

INTERVENTIONS:
Procedure: Superficial Parasternal Block (SIPB) — Immediately after induction of general anesthesia, ropivacaine 0.5% with dexamethasone 8mg/20ml (maximum dose 1.5 mg/kg ropivacaine per each side) is administered in the superficial parasternal intercostal plane using real-time ultrasound guidance.
  Arms: SUPERFICIAL PARASTERNAL INTERCOSTAL PLANE BLOCK (SPIPB)
Procedure: Erector Spinae Plane Block (ESPB) — Immediately after induction of general anesthesia, ropivacaine 0.5% with dexamethasone 8mg/20ml (maximum dose 1.5 mg/kg ropivacaine per each side) is administered in the plane deep to the erector spinae muscle, typically at the level of the 5th thoracic vertebra, under real-time ultrasound guidance.
  Arms: ERECTOR SPINAE PLANE BLOCK (ESPB)
Drug: General anesthetic — During general anesthesia, fentanyl is administered according to NOL monitoring.
  Other Names: NOL-directed general anesthesia
Drug: Morphine — Morphine 0.03 mg/kg is administered postoperatively for NRS scores equal or higher than 4.
  Other Names: Postoperative analgesia

SUMMARY:
This clinical trial focuses on an elaborate, propensity-matched, non-inferiority comparison of NOL-guided Superficial Parasternal Intercostal Plane Block (SPIPB) and Erector Spinae Plane Block (ESPB) within the context of open-heart surgery with cardiopulmonary bypass.

DETAILED DESCRIPTION:
A. Ethics

Local Ethics Committee approval and Informed Consent from patient or next-of-kin are obtained prior to study enrollment.

B. Study enrollment

Forty consecutive adult patients scheduled for elective open cardiac surgery under general anesthesia are to receive general anesthesia plus SPIPB. This prospective group of patients will be matched one-to-one to a historical group of 55 patients that underwent open cardiac surgery under general anesthesia combined with ESPB.

C. Methods

C1. Preinduction

* 16-G peripheral intravenous cannula and radial artery catheter.
* Five-lead ECG, pulse oximetry, non-invasive and invasive blood pressure monitoring.
* Analgesia monitor - the NoL index (PMD200TM, Medasense) finger probe will be connected to the index finger of the non-cannulated hand.
* Surgical antibiotic prophylaxis (Cefuroxime 1.5g).
* Stress ulcer prophylaxis (omeprazole 40 mg).

C2. Superficial Parasternal Intercostal Plane Block (SPIPB)

After induction, skin asepsis with chlorhexidine 2% is performed on the anterior chest wall. A high-frequency linear ultrasound probe is positioned parasagittally, 2 cm from midline, bilaterally, at the level of the 4th rib. A 25-G echogenic block needle is inserted at a 20⁰-30⁰ angle in a caudal-to-cephalad direction until the tip of the needle reaches the interfascial plane between the pectoralis major muscle and the internal intercostal muscle. Correct hydrodissection is first certified using normal saline. Subsequently, ropivacaine 0.5% with dexamethasone 8mg/20ml is used and maximum spread is attained by slowly advancing the needle as the interfascial plane splits up ahead. A maximum dose of 3mg/kg ropivacaine is used, corresponding to 1.5 mg/kg per side (e.g., 20 ml ropivacaine 0.5% / side for a 70kg adult).

C3. General anaesthesia

Monitoring

* End tidal CO2 (ETCO2).
* Bispectral index (BIS) monitoring (target 40-60).
* The nociception monitor (PMD200TM, Medasense) is started before induction.
* CVP insertion into the right internal jugular vein under ultrasound guidance.
* Urinary catheter, rectal temperature probe placement.

Induction

* Propofol 1-1.5 mg/kg or Etomidate 0.2-0.3 mg/kg.
* Fentanyl 5 mcg/kg.
* Atracurium 0.5 mg/kg.

Maintenance of anaesthesia

* Sevoflurane in O2 during periods of preserved pulmonary blood flow and mechanical ventilation.
* Propofol infusion during periods of extracorporeal support.
* Atracurium 0.2-0.3 mg/kg/h for adequate neuromuscular blockade.

Analgesia

1. Analgesic drugs

   * Fentanyl: bolus 1.5 mcg/kg.
   * Paracetamol: 1-gram following induction of general anaesthesia.
2. Analgesia monitoring

   * NoL index provides a multiderivative assessment of nociception before cardiopulmonary bypass (CPB) initiation. Optimal analgesia is defined as a NoL index of 10-25.
   * Mean arterial blood pressure (MAP) provides post-CPB decision loop: targets are within ± 15% of MAP recorded during optimum NOL.

C4. Postoperative

Extubation criteria

* Normothermia (T◦ ≥ 36◦C).
* No clinical bleeding.
* Wakefulness.
* Hemodynamic stability (MAP ≥ 60 mmHg and lactate ≤ 2 mmol/L) with minimal vasoactive support (dobutamine < 5 µg/kg/min and norepinephrine < 100 ng/kg/min).
* Adequate gas exchange:
* Tidal volume ≥ 5 ml/kg.
* Adequate airway reflex to handle secretions.

Analgesia

* Paracetamol 1g iv every 6 hours.
* Morphine bolus 0.03 mg/kg for NRS > 3.

ELIGIBILITY:
Inclusion Criteria:

1. Informed Consent.
2. Elective heart surgery with sternotomy and bypass.
3. Hemodynamic stability prior to induction.
4. Sinus rhythm.

Exclusion Criteria:

1. Known allergy to any of the medications used in the study.
2. BMI > 35.
3. Patient refusal to participate in the study.
4. Coagulopathy (INR > 1.5, APTT > 45, Fibrinogen < 150 mg/dl).
5. Non-elective/emergent and/or redo surgery.
6. ASA ≥ 4.
7. Any preoperative hemodynamic support (mechanical or pharmaceutical).
8. Severe LV dysfunction (LVEF ≤ 30%).
9. Severe RV dysfunction.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Fentanyl consumption (µg/kg) | during intraoperative period
  Intraoperative opioid consumption after goal directed monitoring of nociception with the NOL index
Morphine consumption (µg/kg) | 48 hours after surgery
  Postoperative opioid consumption

SECONDARY OUTCOMES:
Quality of postoperative analgesia | 6 hours, 12 hours, 24 hours and 48 hours after extubation/ICU admission and 1 hour after drain removal
  Assessment - numerical rating scale (NRS) (minimum of 0, maximum of 10)
Time to extubation | up to 24 hours after surgery
  Following ICU admission, the time it takes to extubate the patient safely
Norepinephrine dose (mcg/kg) | intraoperative, 6 hours and 12 hours after surgery
  Cumulative dose of Norepinephrine
Time to weaning-off norepinephrine | up to 96 hours after surgery
  Following ICU admission, the time it takes to stop norepinephrine administration
Dobutamine dose (mcg/kg) | intraoperative, 6 hours and 12 hours after surgery
  Cumulative dose of Dobutamine
Time to first dose of morphine | any time for 48 hours
  Following admission, the time it takes a patient to request morphine rescue analgesia
Extubated patients | 2 hours after surgery
  Number of extubated patients after ICU admission
Norepinephrine-free patients | 2 hours after surgery
  Number of patients without norepinephrine support
Morphine-free patients | 48 hours after surgery
  Number of patients who did not require morphine rescue analgesia

CONTACTS AND LOCATIONS:
Overall Officials: Serban-Ion Bubenek-Turconi, Professor, Study Director — "Prof CC Iliescu" Emergency Institue for Cardiovascular Diseases
Locations (1):
- Cosmin Balan, Bucharest, Sector 2, Romania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Balan C, Tomescu DR, Valeanu L, Morosanu B, Stanculea I, Coman A, Stoian A, Bubenek-Turconi SI. Nociception Level Index-Directed Erector Spinae Plane Block in Open Heart Surgery: A Randomized Controlled Clinical Trial. Medicina (Kaunas). 2022 Oct 16;58(10):1462. doi: 10.3390/medicina58101462. PMID 36295622
- [Result] Balan C, Tomescu DR, Bubenek-Turconi SI. Nociception Control of Bilateral Single-Shot Erector Spinae Plane Block Compared to No Block in Open Heart Surgery-A Post Hoc Analysis of the NESP Randomized Controlled Clinical Trial. Medicina (Kaunas). 2023 Jan 30;59(2):265. doi: 10.3390/medicina59020265. PMID 36837467